CLINICAL TRIAL: NCT03630614
Title: A Randomized, Placebo Controlled, Double Blind, Double Dummy, Multicenter Trial Comparing Electronic Cigarettes With Nicotine to Varenicline and to Electronic Cigarettes Without Nicotine.
Brief Title: Randomized Trial of Electronic Cigarettes With or Without Nicotine in Smoking Cessation.
Acronym: ECSMOKE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P150952J; 2017-003588-37 (EudraCT Number)
Record Dates: First submitted 2018-07-09; First posted 2018-08-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation; Smoking, Cigarette; Electronic Cigarette
Keywords: smokers; electronic cigarette; nicotine; varenicline; randomized; double blind; double dummy
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking; Vaping | interventions — Electronic Nicotine Delivery Systems; Nicotine; Varenicline

STUDY DESIGN:
Intervention Model Description: Randomized, placebo and reference treatment controlled, multicenter, double blind, double dummy, parallel group, pivotal, phase III trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electronic cigarette condition (Experimental): Electronic cigarette with nicotine (ECwN) plus placebo tablets of varenicline
  Interventions: Drug: Electronic cigarette with nicotine (ECwN) plus placebo tablets of varenicline
- Varenicline condition (Active Comparator): Reference group: Electronic cigarette without nicotine (ECwoN) plus active varenicline tablets
  Interventions: Drug: Electronic cigarette without nicotine (ECwN) plus active varenicline tablets
- Placebo condition (Placebo Comparator): Electronic cigarette without nicotine (ECwoN) plus placebo tablets of varenicline
  Interventions: Drug: Electronic cigarette without nicotine (ECwoN) plus placebo tablets of varenicline

INTERVENTIONS:
Drug: Electronic cigarette without nicotine (ECwN) plus active varenicline tablets — The ECwN group use EC liquids containing 0 mg/mL of nicotine. Because nicotine delivery can be adjusted according to the user's need, all participants are able to adjust their individual nicotine dose by varying the wattage of their EC, by varying puff frequency and puff volume similarly as they are doing (or used to do) with conventional cigarettes.
  EC device:
  Mini iStick kit (20 W) Eleaf Clearomiser :GS Air M with resistance of 1.5 ohm, the clearomiser's Pyrex window is of blue colour not allowing to distinguish an eventual coloration of the e-liquid containing nicotine. Liquids for EC use are delivered in white opaque 10 mL vials not allowing to distinguish the color of the liquid.
  Varenicline, Champix® 0.50 mg tablets Posology of vareniclin follows varenicline's monograph.
  Other Names: Vareniclin condition
  Arms: Varenicline condition
Drug: Electronic cigarette without nicotine (ECwoN) plus placebo tablets of varenicline — The ECwoN group receives EC liquids with 0 mg/mL of nicotine on a double blind manner (in identical non-transparent refill bottles of 10 mL).
  Placebo of varenciline The placebo of varenicline is presented as a capsular-shaped, biconvex, white film-coated tablet. Posology of varenicline or its placebo follows varenicline's monograph.
  Other Names: Placebo condition
  Arms: Placebo condition
Drug: Electronic cigarette with nicotine (ECwN) plus placebo tablets of varenicline — The ECwN group use EC liquids containing 12 mg/mL of nicotine. Placebo of varenciline The placebo of varenicline is presented as a capsular-shaped, biconvex, white film-coated tablet. Posology of varenicline or its placebo follows varenicline's monograph.
  Other Names: Electronic cigarette condition
  Arms: Electronic cigarette condition

SUMMARY:
Background:

Electronic cigarettes (EC) mainly containing nicotine (88-95 % of users) are widely and growingly used worldwide. It is estimated that there were 1.7 million daily users in France in 2016. Although the number of publications about its use is increasing exponentially, there are no evidence based, unbiased, head-to-head comparison data about its efficacy as an aid to smoking cessation. As of today, only two head-to-head randomized studies have been published, both reported negative results at the main endpoint but they used first and second generation EC delivering nicotine with low or unknown bioavailability. Recent EC deliver nicotine with largely improved bioavailability.

One of the randomized studies compared EC with and without nicotine to nicotine patch and reported similar smoking cessation rate at main outcome. However, there is no published, double blind study comparing EC use with a well-studied, licensed smoking cessation medication.

Superiority of EC with nicotine compared to EC without nicotine and to a reference smoking cessation medication while collecting also straightforward information about safety, would allow proposing EC with nicotine to the large population of smokers who intend to quit and situate it among the approved smoking cessation treatments.

The clinical study's hypothesis:

EC containing nicotine can be considered as a nicotine replacement therapy having, probably, a better bioavailability of nicotine than the marketed pharmaceutical NRTs, first line medications of smoking cessation. It is therefore of interest to compare EC containing nicotine to EC without nicotine but also to a reference medication with demonstrated efficacy in smoking cessation. We hypothesize that EC with nicotine provides a higher smoking abstinence rate than EC without nicotine and may be as good as varenicline, our reference medication.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, multicenter, double dummy, parallel groups, phase III type pivotal trial.

Included participants are randomly assigned to one of the 3 groups:

A) Control group: Electronic cigarette without nicotine (ECwoN) plus placebo tablets of varenicline: placebo condition B) Experimental group: Electronic cigarette with nicotine (ECwN) plus placebo tablets of varenicline: ECwN condition C) Reference group: ECwoN plus varenicline tablets: varenicline condition Ratio: A:B:C= 1:3:3 Each participant uses an EC and 2x2 tablets per day. Group allocation is stratified by age at cut off of 45 years.

Enrolment is initiated by two ways:

• Potential participants aware of the study register at the study's recruitment website; call in or send an email followed by a phone screen. The screening starts with the participant's information about the study's aims, constraints, benefits and risks. A maximum one week delay of reflection is allowed if the potential participant is asking for a delay to sign his/her consent form.

After screening, an appointment for the inclusion visit is provided at the closest investigation center.

• Referred or self-referred potential participants consulting for smoking cessation are proposed an inclusion visit.

The participant is informed that in this study, the smoking cessation shall occur within 15 days following the signature of the written consent.

Baseline visit = inclusion visit = V0 The Inclusion visit can immediately follow the screening visit if the participant does not need time for reflection.

The investigator checks the inclusion and exclusion criteria and if the participant is conform to them, the investigator collects informed written consent from the participant and he/she is included in the trial. The randomization can immediately follow the inclusion.

A target quit date (TQD) is defined together with the participant. The TQD defines the date when the randomized participant stops smoking. This is the starting date of the post-quit period. Start of treatment should occur within 7 days after the randomization visit.

All treatments are launched one week before the TQD. During this period smoking conventional cigarettes is allowed.

Follow-up visits : Visit 1 to Visit 6 Target quit date (TQD) should occur between 7 and 15 days after randomization. The first post-quit date visit (Visit 1)is at Week 2 after TQD i.e. 3 weeks after treatment initiation = Day 21 after treatment initiation.

Visit 2 is at Week 4 after TQD i.e. 5 weeks after treatment initiation = Day 35 after treatment initiation.

Visit 3 is at Week 8 after TQD i.e. 9 weeks after treatment initiation = Day 63 after treatment initiation.

Visit 4 is at Week 10 after TQD i.e. 11 weeks after treatment initiation = Day 77 after treatment initiation.

Visit 5 is at Week 12 after TQD i.e. 13 weeks after treatment initiation = Day 91 after treatment initiation.

Visit 6 is at Week 24 after TQD i.e. 25 weeks after treatment initiation = Day 175 after treatment initiation.

The visits should be realized +/- 5 days with respect to the planned date of the visits.

End of study visit The end of research visit is the Visit 6, at week 24 after TQD. This visit is identical to the previous follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Smokers smoking at least 10 cigarettes/day (factory made or roll-your-own) in the past year
2. Aged 18 to 70 years
3. Motivated to quit defined as a score > 5 on a visual rating scale ranging from 0 (not motivated at all) to 10 (extremely motivated)
4. Signed written informed consent
5. Understanding and speaking French
6. Women of childbearing age can be included if they use an effective contraceptive method: either hormonal contraception or an intrauterine device started at least one month before the first research visit
7. Individual affiliated to a health insurance system as defined by the sponsor (except Aide Médicale d'État =AME)
8. Previous failure of nicotine replacement therapy for smoking cessation

Exclusion Criteria:

1. any unstable disease condition within the last 3 months defined by the investigator as major change in symptoms or treatments such as 1.1.recent myocardial infarction, 1.2.unstable or worsening angina 1.3.severe cardiac arrhythmia 1.4.unstable or uncontrolled arterial hypertension 1.5.recent stroke 1.6.cerebrovascular disease 1.7.obliterative peripheral arterial disease 1.8.cardiac insufficiency 1.9.diabetes 1.10.hyperthyroidism 1.11.pheochromocytoma 1.12.severe hepatic insufficiency 1.13.history of seizures 1.14.severe depression 1.15.chronic obstructive pulmonary disease (COPD)
2. any life threatening condition with life-expectancy of less than 3 months
3. alcohol use disorder defined as a score ≥ 10 on the AUDIT-C questionnaire
4. abuse of or dependence on illegal drugs in the last 6 months revealed by the medical history
5. regular use of tobacco products other than cigarettes
6. current or previous (last 6 months) use of electronic cigarette
7. pregnant women
8. breastfeeding women
9. protected adults
10. current or past 3 months participation in another interventional research
11. current or past (last 3 months) use of smoking cessation medication such as varenicline, bupropion, nicotine replacement therapies
12. known lactose intolerance (placebo tablets contain lactose)
13. hypersensitivity to the active substance or to any of the excipients
14. known severe renal failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2018-10-17 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Continuous smoking abstinence rate | Weeks 9 to 12
  Abstinence from conventional/combustible cigarettes during the last 4 weeks (weeks 9 to 12) of the treatment period of 3 months defined at Visit 4 AND Visit 5 as self-report of no smoking during the previous 2 weeks confirmed by expired air CO ≤ 8 ppm.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | From randomisation up to end of study (Week 24 after target quit date).
  The safety profile of electronic cigarette with nicotine comparatively to electronic cigarettes without nicotine and varenicline
Point prevalence abstinence rate: 7-day smoking abstinence at each visit. | From randomisation up to end of study (Week 24 after target quit date).
Time to relapse to smoking after the predefined quit day. | From randomisation up to end of study (Week 24 after target quit date).
Change in cigarettes/day consumption | From randomisation up to end of study (Week 24 after target quit date).
French Tobacco Craving Questionnaire of 12 items (FTCQ-12) | From randomisation up to end of study (Week 24 after target quit date).
  Change in craving for tobacco
Minnesota Nicotine Withdrawal Scale | From randomisation up to end of study (Week 24 after target quit date).
  Change in tobacco withdrawal symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Pitié-Salpétrière, Paris, France

REFERENCES:
- [Derived] Berlin I, Dautzenberg B, Lehmann B, Palmyre J, Liegey E, De Rycke Y, Tubach F. Randomised, placebo-controlled, double-blind, double-dummy, multicentre trial comparing electronic cigarettes with nicotine to varenicline and to electronic cigarettes without nicotine: the ECSMOKE trial protocol. BMJ Open. 2019 May 24;9(5):e028832. doi: 10.1136/bmjopen-2018-028832. PMID 31129603